CLINICAL TRIAL: NCT06285032
Title: Addressing Loneliness in Primary Care Patients on Chronic Opioids to Prevent Opioid Misuse
Brief Title: Decreasing Loneliness to Optimize Pain Care
Acronym: DLoop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sebastian Tong, Assistant Professor: School of Family Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017244; R34DA058325 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Loneliness; Opioid Use
Keywords: Loneliness; Opioid use; Chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy (CBT) (Experimental): Participants will be randomized to the CBT group (N=34). CBT groups will meet for 1 hour via Zoom, for 8 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy (CBT)
- Social Navigation Group (Experimental): Participants will be randomized to the social navigation group (N=34). Social navigation group will meet for 30 mins via Zoom, for 8 weeks.
  Interventions: Behavioral: Social Navigation Group
- Usual Care Group (Experimental): Participants will be randomized to the usual care group (N=34). Participants in this group will resume to their usual standard of care for 8 weeks.
  Interventions: Behavioral: Controlled Group

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy (CBT) — Individuals will participate in a series of eight, 1hour weekly group sessions delivered by a study interventionalist who is a licensed social worker (see personnel list) using a HIPAA-compliant videoconferencing platform (Zoom). Each group will consist of 6-10 participants and participants randomized to this intervention will select between a series of date/time options. The investigators plan to run four groups with staggered start times. All participants will receive digital copies of the workbook for this intervention and each session, they will be given assignments to practice the strategies they learn during the intervention.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Social Navigation Group — Those in the social navigation intervention, will meet with a navigator weekly through a virtual visit (HIPAA-compliant videoconferencing or phone call based on patient preference) over the course of 8 weeks. Each virtual visit will last approximately 30 minutes with a longer initial intake visit lasting 60 minutes. During the intake visit, the navigator will complete a patient narrative and an inventory of the patient's existing social network, former social network and interests. Using this, the navigator will work with the patient to develop an action plan to promote, establish or re-establish social connections. The action plan will be referenced and refined throughout the course of the 8 weeks. They will suggest specific social activities and connect patients to resources such as, community-based organizations or local social groups matched to individual participant interest to assist with social connection
  Arms: Social Navigation Group
Behavioral: Controlled Group — Those randomized to the control group will receive usual care from their primary care clinician. At the conclusion of the study (after the final outcomes are collected), they will be offered a list of possible community-based organizations for social connection.
  Arms: Usual Care Group

SUMMARY:
Loneliness, which is the perceived feeling of insufficient personal relationships, is related to higher risk for inappropriate opioid use and opioid use disorders in patients who are taking opioids long-term. The study seeks to pilot test the evidence-based loneliness interventions of psychological therapy and social navigation in patients on chronic opioids treated in primary care practices to determine if reducing loneliness can lower opioid misuse.

DETAILED DESCRIPTION:
Patients with chronic pain on opioids frequently experience loneliness, which is associated with poorer health outcomes and higher risks for opioid misuse and opioid use disorder. Given that almost half of opioids are prescribed in primary care, a critical need exists for the development and testing of interventions to reduce loneliness in primary care patients at risk for opioid misuse. The long-term goal of the study is to reduce opioid misuse and opioid use disorder by addressing loneliness in primary care with patients on chronic opioids. Interventions addressing maladaptive social cognition through cognitive behavioral therapy and improving social support through social navigation have been shown to be effective in reducing loneliness and improving outcomes in other fields but have not been tested in patients at risk for substance use disorder.

Aims

* To refine both the social navigation and psychological CBT loneliness interventions for patients in primary care on chronic opioids
* To assess the feasibility of implementing a 3-arm pilot randomized clinical effectiveness trial testing a psychological CBT and a social navigation intervention to address loneliness in primary care patients.
* To determine the distribution and variability in the mediating outcome (loneliness), the primary outcome (opioid misuse) and secondary outcomes, including opioid dose, functional status and patient-reported pain outcomes in the pilot randomized clinical effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* On chronic opioids (defined as defined as 3 or more months receiving prescribed opioids [functional definition is 3 or more opioid prescriptions each less than 21 days apart as per our prior studies])
* With a score greater or equal to 6 on the UCLA Loneliness 3-item Scale
* Have a chronic pain diagnosis

Exclusion Criteria:

* Have cancer-related pain
* Are on palliative care or live in a controlled setting (i.e., assisted living, nursing home or inpatient treatment facility)
* Have an upcoming scheduled surgery
* Severe cognitive impairment or active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Opioid Misuse | Baseline, post-intervention (2 weeks after the completion of the intervention), and month 3 after completed intervention.
  The primary outcome is to see changes in opioid misuse, which the investigators will measure using the Current Opioid Misuse Measure (COMM). The investigators will give the COMM at baseline, post-intervention (2 weeks after intervention completion), and 3 months after the intervention has been completed to find out changes in behaviors. Those with a score of 9 or greater are consider positive for misuse (min=0, max score=68).

SECONDARY OUTCOMES:
Determine Functional Outcome | Baseline, post-intervention (2 weeks after the completion of the intervention), and month 3 after completed intervention.
  The investigators will use the Patient Reported Outcomes Measurement Information (PROMIS) pain interference (version 6b) to measure changes in functionality. Investigators will interpret data from the survey and look at participants who indicate any amount of pain (min=0, max score=30). The PROMIS scale is used to track pain interference, especially for those who frequently struggle with chronic pain and therefore, are on chronic opioids.

OTHER OUTCOMES:
Loneliness | Baseline, post-intervention (2 weeks after the completion of the intervention), and month 3 after completed intervention.
  The mediating outcome is to track changes in loneliness using the University of California, Los Angeles Loneliness (UCLA). A score of 6 or higher (max score=80) will indicate participants experience some to severe loneliness. Those with scores of 5 or lower (min=0) indicate that they do not experience loneliness and therefore, will not be considered in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Tong, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Tong ST, Ma KPK, Pleho A, Keiser B, Hsu C, Ehde DM, Curran MC, Tsui JI, Raue PJ, Stephens KA. Comparing cognitive behavioral therapy and social prescribing in patients with loneliness on long-term opioid therapy to reduce opioid misuse: protocol for a randomized controlled trial. Addict Sci Clin Pract. 2024 Sep 11;19(1):66. doi: 10.1186/s13722-024-00498-y. PMID 39261953